CLINICAL TRIAL: NCT05061667
Title: Thoracic Paravertebral Block Versus Rhomboid Block for Postoperative Pain Control in Thoracic Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Koç University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021.066.IRB1.022
Record Dates: First submitted 2021-09-22; First posted 2021-09-29 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2021-05

CONDITIONS: Postoperative Pain
Keywords: Thoracic surgery; Postoperative pain; Rhomboid block; Paravertebral block
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Active Comparator): Group I will consist of randomly assigned patients scheduled for thoracic surgery. These patients will recieve paravertebral block which is already proven to be effective in postoperative pain. After applying standart monitors to the patient and proper positioning in the operating room, paravertebral block will be performed at the planned surgical side using high frequency (8-18 MHz) linear probe of GE Logiq S7 (General Electric Healthcare, Little Chalfont, United Kingdom). 20 ml of 0.25% bupivacaine will be administered into the paravertebral space at T5-T6 vertebra levels using a 50 mm 22 G block needle (BBraun, Melsungen, Germany).
  Interventions: Procedure: Thoracic Paravertebral Block
- Group II (Experimental): Group II will consist of randomly assigned patients scheduled for thoracic surgery. These patients will recieve rhomboid block which is being experimented for its efficacy in postoperative pain. After applying standart monitors to the patient and proper positioning in the operating room, rhomboid block will be performed at the planned surgical side using high frequency (8-18 MHz) linear probe of GE Logiq S7 (General Electric Healthcare, Little Chalfont, United Kingdom). 20 ml of 0.25% bupivacaine will be administered into the plane between rhomboid muscle and intercostal muscles, medial to scapula at T5-T6 vertebra levels using a 50 mm 22 G block needle (BBraun, Melsungen, Germany).
  Interventions: Procedure: Rhomboid Block

INTERVENTIONS:
Procedure: Thoracic Paravertebral Block — Paravertebral block for postoperative analgesia in thoracic surgery
  Other Names: TPVB
  Arms: Group I
Procedure: Rhomboid Block — Rhomboid block for postoperative analgesia in thoracic surgery
  Arms: Group II

SUMMARY:
The main aim of this study is to compare thoracic paravertebral block and rhomboid block for postoperative analgesia and analgesic usage in thoracic surgeries.

DETAILED DESCRIPTION:
Patients with scheduled thoracic surgery are going to be enrolled for this study. Patients will be randomized and separated in two groups. Group I will receive thoracic paravertebral block, group II will receive rhomboid block. Each group will receive patient controlled analgesia with intravenous fentanyl. Patients will be monitored at postoperative 1st, 3rd, 6th, 12th, 24th hours and their VAS scores, adverse reactions like nausea and vomiting, total analgesic usage, additional analgesic need and time of the first report of pain will be filed. Then the two groups will be compared and evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for general thoracic surgery
* ASA I-III

Exclusion Criteria:

* Patients without consent
* Emergency surgeries
* Pregnancy
* Coagulopathies and bleeding diathesis
* Allergy to local anesthetics
* Local skin infection at the puncture site

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
Difference in Visual Analogue Scale (VAS) scores between two groups | 24 hours
  Statistically significant difference in VAS scores at 1st, 3rd, 6th, 12th, 24th hours between two groups. On a scale of 0 to 10, where 0 means no pain and 10 means the worst imaginable pain.
Difference in additional analgesic usage between two groups | 24 hours
  Intravenous patient controlled analgesia usage and additional analgesic dosages will be filed as miligrams or micrograms at 1st, 3rd, 6th, 12th, 24th hours.

SECONDARY OUTCOMES:
Incidence of nausea and vomiting | 24 hours
  Incidence of symptoms like nausea and vomiting will be filed at 1st, 3rd, 6th, 12th, 24th hours. On a scale of 0 to 1, where 0 means no symptoms and 1 means nausea and vomiting.
Patient satisfaction | 24 hours
  Patient will be reevaluated at 24th hour for analgesic satisfaction. On a scale of 0 to 3, where 0 means not satisfied and 3 means satisfied.

CONTACTS AND LOCATIONS:
Locations (1):
- Koç University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Data collected for the study, including de-identified individual participant data will be made available to other within 6 months after the publication of this trial, as will additional related documents (study protocol, statistical analysis plan and informed consent form), for academic purposes (e.g., meta-analyses), upon request to the corresponding author, and with a signed data access agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 6 months after the publication
Access Criteria: Academic purposes

REFERENCES:
- [Background] Ciftci B, Ekinci M, Atalay YO. Ultrasound-guided rhomboid intercostal block provides effective pain control after video-assisted thoracoscopic surgery: a brief report of three cases. Korean J Anesthesiol. 2021 Aug;74(4):355-357. doi: 10.4097/kja.20538. Epub 2020 Nov 17. No abstract available. PMID 33198430
- [Background] Longo F, Piliego C, Martuscelli M, Tomaselli E, Crucitti P, Longo F, Agro FE. Rhomboid intercostal and subserratus plane block for intubated uniportal video-assisted thoracoscopic surgery lobectomy. J Clin Anesth. 2020 Oct;65:109881. doi: 10.1016/j.jclinane.2020.109881. Epub 2020 May 26. No abstract available. PMID 32470838
- [Background] Longo F, Piliego C. Rhomboid intercostal and subserratus plane block for non-intubated video-assisted thoracoscopic surgery. J Clin Anesth. 2020 May;61:109612. doi: 10.1016/j.jclinane.2019.09.006. Epub 2019 Oct 24. No abstract available. PMID 31668692